CLINICAL TRIAL: NCT02876887
Title: Cocoa to Improve Walking Performance in Peripheral Artery Disease
Acronym: COCOA-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00202741; R21AG050897 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-08-24 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocoa (Active Comparator): Three servings per day of epicatechin-rich (75 mg daily) cocoa beverages for six months.
  Interventions: Drug: Cocoa
- Placebo (Placebo Comparator): Three servings per day of placebo beverages for six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cocoa
  Arms: Cocoa
Drug: Placebo
  Arms: Placebo

SUMMARY:
The COCOA-PAD trial will determine whether epicatechin-rich cocoa daily for six months improves walking performance in individuals with peripheral artery disease compared to placebo.

DETAILED DESCRIPTION:
Therapeutic properties that target pathophysiologic impairments in PAD. These therapeutic properties include improved skeletal muscle mitochondrial function, increased skeletal muscle capillary density, and favorable changes in skeletal muscle levels of myostatin and follistatin that increase muscle mass and strength. Cocoa also protects against ischemia-reperfusion injury, improves endothelial function, and reduces oxidative stress. In summary, epicatechin-rich cocoa targets and reverses several pathophysiologic processes that are common in PAD and that are associated with functional impairment and functional decline in PAD. However, the effect of chronic daily cocoa consumption on functional decline has not been studied in older people with PAD.

The COCOA-PAD trial is a pilot study of 44 PAD participants age 60 and older: a double-blind, randomized controlled pilot clinical trial to provide preliminary data to address the hypothesis that chronic daily epicatechin-rich cocoa improves lower extremity functioning in older people with PAD by improving mitochondrial oxidative metabolism, increasing calf muscle capillary density, promoting calf skeletal muscle mitochondrial biogenesis, and improving endothelial function.

In the primary aim, the investigators will determine whether PAD participants randomized to an epicatechin-rich cocoa beverage have greater increases or smaller declines in six-minute walk performance at 6-month follow-up, compared to those randomized to an identical appearing placebo drink with comparable caloric composition. In the secondary aims, the investigators will determine whether PAD participants randomized to cocoa have improved treadmill walking performance, improved brachial artery flow-mediated dilation, favorable changes in calf muscle biopsy measures of mitochondrial function, mitochondrial biogenesis, follistatin, myostatin, and capillary density, increased calf skeletal muscle regeneration and reduced oxidative stress, and increased MRI-measured calf muscle perfusion. Outcome measures will be carefully timed relative to the last intervention dose to distinguish between the acute vs. chronic effects of cocoa-epicatechin.

If the hypotheses are correct, results will be used to design a large, definitive randomized controlled trial of epicatechin-rich cocoa to improve lower extremity functioning and prevent mobility loss in the large and growing number of older people who are disabled by PAD.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be age 60 and older.
2. All participants will have PAD. PAD will be defined as follows. First, an ABI < 0.90 at baseline is an inclusion criterion for PAD. Second, potential participants with an ABI > 0.90 who have vascular lab evidence of PAD or angiographic evidence of PAD will be eligible.

Exclusion Criteria:

1. Above- or below-knee amputation.
2. Critical limb ischemia.
3. Wheelchair-bound or requiring a cane or walker to ambulate.
4. Walking is limited by a symptom other than PAD.
5. Baseline six-minute walk value of <500 feet or >1,600 feet
6. Lower extremity revascularization, major orthopedic surgery, cardiovascular event, or coronary revascularization in the previous three months.
7. Planned revascularization or major surgery during the next six months.
8. Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who require oxygen only at night may still qualify.]
9. Mini-Mental Status Examination (MMSE) score < 23 or dementia.
10. Unwilling to attend three visits in one week for final outcome measures.
11. Allergy to chocolate.
12. Unwilling or unable to consume products manufactured on the same equipment that processes peanuts, tree nuts, egg, wheat, soy, and milk.
13. Use of cocoa-containing dietary supplements.
14. Unwilling to give up major dietary sources of epicatechin during the study.
15. Symptoms of heart failure or angina that limit walking activity more than ischemic leg symptoms, increase in angina, or angia at rest (i.e. unstable angina).
16. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
17. Non-English speaking, a visual impairment that limits walking ability.
18. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDermott MM, Criqui MH, Domanchuk K, Ferrucci L, Guralnik JM, Kibbe MR, Kosmac K, Kramer CM, Leeuwenburgh C, Li L, Lloyd-Jones D, Peterson CA, Polonsky TS, Stein JH, Sufit R, Van Horn L, Villarreal F, Zhang D, Zhao L, Tian L. Cocoa to Improve Walking Performance in Older People With Peripheral Artery Disease: The COCOA-PAD Pilot Randomized Clinical Trial. Circ Res. 2020 Feb 28;126(5):589-599. doi: 10.1161/CIRCRESAHA.119.315600. Epub 2020 Feb 14. PMID 32078436

RESULTS

PARTICIPANT FLOW:
Groups:
- Cocoa: Three servings per day of epicatechin-rich (75 mg daily) cocoa beverages for six months.
  Cocoa
- Placebo: Three servings per day of placebo beverages for six months.
  Placebo
Period: Overall Study
Arm/Group | Cocoa | Placebo
Started | 23 | 21
Completed | 19 | 21
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocoa | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 73 (7) | 72 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 12 | 31
  White | 4 | 9 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six-minute Walk Distance
Description: Following a standardized protocol, participants walked up and down a 100-ft hallway for 6 minutes after instruction to cover as much distance as possible.
Time Frame: Change from baseline to six-month follow-up. Note - There will be two measures: One 2-3 hours after the final study beverage dose and one 24 hours after the final dose.
Population: Nineteen and 21 study participants in the cocoa and placebo groups, respectively, completed the six-minute walk at both baseline and 6-month follow-up.
Measure: Mean (90% Confidence Interval); unit: meters
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 19 | 21
meters
  Six-month, 2.5 hours after study beverage (meters) | 18.4 [0.34 to 36.5] | -24.2 [-40.7 to -7.8]
  Six-month, 24 hours after study beverage (meters) | 15.1 [-1.9 to 32.1] | -2.9 [-19.4 to 13.6]

2. Secondary Outcome: Change From Baseline in Maximal and Pain-free Treadmill Walking Time
Description: Maximal treadmill walking time and time to ischemic leg symptom onset were measured using the Gardner-Skinner protocol at baseline and 6-month follow-up.
Time Frame: Change from baseline to six-month follow-up
Population: Eighteen and 19 study participants in the cocoa and placebo groups, respectively, participated in both the baseline and 6-month follow-up treadmill test.
Measure: Mean (90% Confidence Interval); unit: minutes
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 18 | 19
minutes
  Maximal treadmill minutes, 48 hrs post beverage | -0.03 [-1.16 to 1.10] | 0.28 [-0.79 to 1.34]
  Pain-free treadmill minutes, 48 hrs post beverage | -0.07 [-1.13 to 1.00] | 0.39 [-0.64 to 1.43]

3. Secondary Outcome: Change in Baseline From Brachial Artery Flow-mediated Dilation: Change in Brachial Artery Diameter
Description: Brachial artery flow-mediated dilation was measured in the proximal brachial artery (B mode and Doppler) after a 12-hour fast by Registered Diagnostic Cardiac Sonographers using a linear array vascular ultrasound transducer (Sequoia Model #256; frequency, 8 MHz; range, 5-8 MHz; Siemens Medical Solutions). A cuff proximal to the visualized brachial artery segment was inflated for 4 minutes at 50 mmHg above systolic pressure. Brachial artery images were obtained 60 seconds after cuff deflation and interpreted by a single reader, blinded to group assignment, at the University of Wisconsin Atherosclerosis Imaging Research Program Core Laboratory. Change in brachial artery diameter will be reported in percent change.
Time Frame: Change from baseline to six-month follow-up. Note - there will be two measures: One 2-3 hours after the final study beverage dose and one 24 hours after the final study beverage dose.
Population: Fifteen and 17 study participants in the cocoa and placebo groups, respectively, participated in brachial artery flow-mediated dilation at baseline and 6-month follow-up.
Measure: Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 15 | 17
Percent change
  FMD change, 2.5 hours after study beverage | -0.65 [-2.08 to 0.78] | 0.63 [-0.69 to 1.96]
  FMD change, 24 hours after study beverage | 0.04 [-1.23 to 1.32] | -0.59 [-1.96 to 0.79]

4. Secondary Outcome: Change From Baseline Accelerometer-measured Physical Activity
Description: Free-living physical activity was acquired over 7 days with the ActiGraph accelerometer. The accelerometer was worn on the right hip and removed only for bathing or sleeping.
Time Frame: Change from baseline to six-month follow-up
Population: Fifteen and 19 study participants in the cocoa and placebo groups, respectively, wore an ActiGraph accelerometer at baseline and 6-month follow-up.
Measure: Mean (90% Confidence Interval); unit: activity counts
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 15 | 19
activity counts | -1919 [-17743 to 13904] | -8981 [-22743 to 4780]

5. Secondary Outcome: Change in Baseline Calf Skeletal Muscle Measures: Abundance of PGC1α, Myostatin and Follistatin
Description: An open-muscle biopsy at baseline was performed in the medial head of the gastrocnemius muscle. Anesthesia was achieved with subcutaneous lidocaine. Subcutaneous tissue was dissected, and ≈250 mg of muscle was removed and immediately prepared for freezing at -80°C. At 6-month follow-up, the biopsy was repeated, adjacent to the original biopsy, identifiable by the scar.
Time Frame: Change from baseline to six-month follow-up
Population: Ten and 6 study participants in the cocoa and placebo groups, respectively, completed muscle biopsy at baseline and 6-month follow-up.
Measure: Mean (90% Confidence Interval); unit: Arbitrary units
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 10 | 6
Arbitrary units
  Abundance of PGC1α | 0.09 [-0.09 to 0.28] | 0.04 [-0.21 to 0.29]
  Abundance of myostatin | 0.26 [0.05 to 0.47] | 0.15 [-0.14 to 0.43]
  Abundance of follistatin | -0.03 [-0.20 to 0.15] | 0.09 [-0.15 to 0.34]

6. Secondary Outcome: Change in Baseline MRI-Measured Calf Skeletal Muscle Perfusion
Description: Arterial spin labeling with cardiovascular magnetic resonance imaging was used to measure changes in calf perfusion at 3 T between PAD participants receiving cocoa versus placebo. A thigh cuff was inflated to 250 mm Hg in the leg with the lowest ABI and rapidly deflated after 5 minutes. Seven control-tagged image pairs were acquired over 60 seconds using pulsed arterial spin labeling pulse sequence with single-shot echo-planar imaging readouts ( eld of view, 200×200 mm; matrix, 64×64; repetition time, 4000 ms; echo time, 32 ms; slice thickness, 10 mm). Perfusion was measured and quantified on a Siemens Healthcare workstation by coinvestigator C.M.K.
Time Frame: Change from baseline to six-month follow-up
Population: Thirteen and 13 study participants in the cocoa and placebo groups, respectively, completed MRI testing at baseline and 6-month follow-up.
Measure: Mean (90% Confidence Interval); unit: ml/min/100 gram
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 13 | 13
ml/min/100 gram | 0.10 [-0.25 to 0.45] | -0.32 [-0.67 to 0.03]

7. Secondary Outcome: Change in Baseline Calf Skeletal Muscle Measures: Citrate Synthase and COX Activity
Description: as for outcome 5
Time Frame: Change from baseline to six-month follow-up
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: (nmol/min/mg protein)
Arm/Group | Cocoa | Placebo
Number analyzed (Participants) | 10 | 6
(nmol/min/mg protein)
  Citrate synthase activity | -0.25 [-3.85 to 3.36] | -1.10 [-5.98 to 3.77]
  COX activity | -4.6 [-37.2 to 28] | -90 [-134.1 to -46]

ADVERSE EVENTS:
Time Frame: Participants were formally asked once per month (1 mo, 2 mo, 3 mo, 4 mo, 5 mo, 6 mo) whether or not they had any hospitalizations.
Description: The following categories were used to define serious adverse events-
  1. Death
  2. Cardiovascular events associated with hospitalization
  3. Hospitalizations for operations or medical conditions other than cardiovascular events.
  4. An untoward medical occurrence resulting in persistent or significant disability/incapacity.
  5. Excessive weight gain in the amount of 20 pounds or more.
  Information regarding other adverse events was not collected.
Arm/Group | Cocoa | Placebo
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 7/23 | 2/21
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cocoa (N=23) | Placebo (N=21)
Hospitalization for depression (Psychiatric disorders) | 1 | 0
Death (Cardiac disorders) | 1 | 0 — Hospitalization for shortness of breath and subsequent heart attack and death.
Lower extremity revascularization (Vascular disorders) | 1 | 0 — Hospitalization for right lower extremity bypass surgery.
Food ulcer with cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 — Hospitalization for infection on his foot. Participant received IV antibiotics and was discharged to a nursing home for subsequent IV antibiotic therapy.
Prostatic enlargement with associated symptoms (Renal and urinary disorders) | 1 | 0 — Hospitalization for symptoms from an enlarged prostate
Other/unknown (Vascular disorders) | 1 | 0 — Hospitalization for acute occlusion of the right femoral artery. She underwent thrombectomy and thrombolysis.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hospitalized for difficulty breathing and swollen ankles, possibly caused by atrial fibrillation or centrilobular emphysema.
Ischemic stroke (Vascular disorders) | 1 | 0 — Hospitalization for ischemic stroke.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hospitalization for coughing and pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT02876887/Prot_SAP_000.pdf